CLINICAL TRIAL: NCT00550875
Title: A Randomised Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Sublingual Immunotherapy With a Depigmented and Polymerized Grass Pollen Extracts in Patients Suffering From Allergic Rhinoconjunctivitis.
Brief Title: Efficacy-safety Study of Sublingual Immunotherapy With Depigmented-polymerized Pollen Extracts to Treat Rhinoconjunctivitis
Acronym: GPIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: María José Gómez, Laboratorios LETI S.L.Unipersonal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6078-PG-OSL-137
Record Dates: First submitted 2007-08-22; First posted 2007-10-30 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergic rhinoconjunctivitis,; Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Biological: Grass pollen allergenic extract (L. perenne-C. dactylon )
- 2 (Experimental): 10* concentration of arm 1
  Interventions: Biological: Grass pollen allergenic extract (L. perenne-C. dactylon )
- 3 (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Grass pollen allergenic extract (L. perenne-C. dactylon ) — Sublingual. 2 drops/daily 1000 DPP/ml 2 years
  Arms: 1
Biological: Grass pollen allergenic extract (L. perenne-C. dactylon ) — Sublingual. 2 drops/daily 10000 DPP/ml 2 years
  Arms: 2
Biological: placebo — Sublingual. 2 drops/daily 2 years
  Arms: 3

SUMMARY:
As the principal objective of this study is to evaluate the efficacy and safety of the treatment measuring the changes in a symptom score, the patient will be asked to fill in a patient diary. This diary will evaluate the week before the patient comes back to receive the treatment. Nose (sneeze, blockage and running), eye (itching, redness and swelling) and chest (breathlessness, wheeze, chest tightness), are scored on a scale from The patient will be instructed to daily assess each one of the symptoms, recording them on an individual symptoms follow-up diary.

DETAILED DESCRIPTION:
The study drug is a sublingual immunotherapy (vaccine) with allergenic extract of grass pollen (Lolium perenne (50%) + Cynodon dactylon (50%)). Sublingual immunotherapy has been available on the European market to treat patients with allergic rhinoconjunctivitis (itching, sneezing, stuffy nose, runny nose) for many years. In this study it will be used as drops under the tongue. At the beginning of the study, you will be given a card that documents that you are taking part. Please carry this with you at all times, in case treatment is necessary at another location. The drops will be given at two doses. The drops are held under the tongue for 2 minutes prior to swallowing.Sublingual Immunotherapy has been shown to be safe and effective in reducing the symptoms of allergic rhinoconjunctivitis (nasal allergy and allergy of the eyes).

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of allergic rhinoconjunctivitis and/or asthma due to hypersensitivity to grass mix Lolium perenne and Cynodon dactylon.
* Male or female subjects between 18 and 50 years old
* Positive skin tests to Lolium perenne and Cynodon dactylon: the wheal produced by the skin test by means of the prick-test technique must be equal or superior to the wheal produced by the positive control of prick test (histamine 10 mg/ml).
* Presence of specific IgE to Lolium perenne and Cynodon dactylon (CAP greater than 17.5K u/L).
* Female subjects must not be sexually active or must be following a medially accepted contraceptive method.
* Pregnancy test negative

Exclusion Criteria:

* Treatment with ß-blocking agents
* Patients suffering from some pathology in which the adrenaline is contraindicated (hyperthyroidism, HTA, cardiopathy, etc.)
* Autoimmune disease (thyroiditis, lupus, etc.)
* Conditions in which the patient can not offer full co-operation, compliance or those with significant psychiatric disturbance.
* Intolerance to aspirin.
* Pregnant women or with pregnancy risk and breast-feeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
AUC for Symptom Score and Mean Symptom Score in the pollen period. | 2 years

SECONDARY OUTCOMES:
Symptom Score, Immunological evaluation,Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ), Adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Potter, PhD, Prof., Principal Investigator — UCT Lung Institute, Cape Town, South Africa
Locations (1):
- Allergy Unit, UCT Lung Institute, Mowbray, Cape Town, South Africa